CLINICAL TRIAL: NCT03839758
Title: Multicenter Randomised Study of Personalized Instrument in Total Shoulder Arthroplasty The P.I.T.S.A. Study
Brief Title: Study of Personalized Instrument in Total Shoulder Arthroplasty The P.I.T.S.A. Study
Acronym: PITSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Dominique Rouleau, Orthopaedic surgeon, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PITSA
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Arthritis
Keywords: Prothesis; Glenoid implantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The evaluator who will perform the follow-up clinical examination will also be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TSA Standard (Active Comparator): This group will include patients schedule for a total shoulder arthroplasty. Glenoid preparation will be done following surgeon evaluation of the 2D CT scan with the institution software. Generic guides included in the regular instrumentation set will be used
  Interventions: Procedure: TSA standard
- RTSA standard (Active Comparator): This group will include patients schedule for a reverse total shoulder arthroplasty. Glenoid preparation will be done following surgeon evaluation of the 2D CT scan with the institution software. Generic guides included in the regular instrumentation set will be used
  Interventions: Procedure: RTSA standard
- TSA blueprint (Experimental): This group will include patients schedule for a total shoulder arthroplasty. Glenoid preparation will be done using the personalized guide provided by Wright-Tornier. This guide will be ordered after CT-scan measurement, using Blueprint software prior to surgery.
  Interventions: Procedure: TSA Blueprint
- RTSA blueprint (Experimental): This group will include patients schedule for a reverse total shoulder arthroplasty. Glenoid preparation will be done using the personalized guide provided by Wright-Tornier. This guide will be ordered after CT-scan measurement, using Blueprint software prior to surgery.
  Interventions: Procedure: RTSA Blueprint

INTERVENTIONS:
Procedure: TSA standard — Glenoid preparation will be done with 2D CT-Scan
  Arms: TSA Standard
Procedure: RTSA standard — Glenoid preparation will be done with 2D CT-Scan
  Arms: RTSA standard
Procedure: TSA Blueprint — Glenoid preparation will be done with Blueprint software
  Arms: TSA blueprint
Procedure: RTSA Blueprint — Glenoid preparation will be done with 2D CT-Scan
  Arms: RTSA blueprint

SUMMARY:
Total shoulder arthroplasty is an effective procedure to improve patients function and to relieve shoulder pain in cases of glenohumeral arthritis. The main challenge of this procedure is implanting the glenoid component. Indeed, surgical exposure is difficult and proper visualization of the glenoid is demanding. The current free-hand method is not precise and especially unreliable in glenoids with severe deformity. Inappropriate reaming and glenoid positioning can cause more bone loss during surgery.

In anatomic prostheses, glenoid component fixation is demanding and is the first component to present loosening at long term follow-up. When it comes to reverse arthroplasty, the glenoid component, once again, requires the most attention. Malpositioning of the glenosphere can cause notching, loosening, and instability.

In order to prevent these complications, precision in glenoid implantation is key. To this end, intraoperative computer navigation would be a helpful tool, but the increased expenses in computer equipment represent massive costs and possibly increases in surgical time. A more affordable option is a personalized guide, for which the only extra expense is the customized guide. These guides are based on precise 3D CT scan templates. Previous studies have evaluated the precision of the guide in vivo and in vitro, but none have measured it in a randomized study. As it represents additional costs, its efficacy needs to be proven before widespread use.

This method may also provide secondary benefits, such as decreasing operating time, lowering short- and long-term complications, and improving efficacy.

The objective of this study is to evaluate the performance of a patient specific glenoid guide.

DETAILED DESCRIPTION:
All participants scheduled for elective primary total shoulder arthroplasty will be contacted by a research assistant. Preoperative status will be characterized by demographic data, range of motion, quality of life, and functional status. A CT Scan and x-rays are part of standard preoperative care and always done prior to total shoulder replacement in our institution; these images will be collected for the study. Patients will be randomized to one of the two groups:

1. Patient-specific glenoid guide group: Glenoid preparation will be done using the personalized guide provided by Wright-Tornier. This guide will be ordered after CT-scan measurement, using Blueprint software prior to surgery.
2. Classic method group: Glenoid preparation will be done following surgeon evaluation of the 2D CT scan with the institution software. Generic guides included in the regular instrumentation set will be used.

The investigators will use the classification proposed by Iannotti et al. to characterize glenoid bone loss prior to surgery. Glenoid bone density will be measured using radiology software (Hounsfield units). Blueprint software will be used to measure the preoperative anatomical characteristics of the glenoid: surface area, version, inclination and subluxation. This will be done prior to surgery in the patient specific group and after surgery in the classic group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with shoulder osteaoarthritis and AVN

Exclusion Criteria:

* Patients with previous shoulder arthroplasty
* Patients with inflammatory arthritis and tumor
* Patients with previous shoulder surgery with metal implant
* Patients refusing 2-year follow-up
* Patients that does not speak English or French
* Patients with current or previous shoulder infection
* Patients with graft during surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Radiological evaluation 1 | 2 weeks post-op
  Comparing the precision of the glenoid implantation during the surgery between both group

SECONDARY OUTCOMES:
Radiological evaluation 2 | 2 years
  Comparaison of the glenoid fixation durong the surgery, between both group
Glenoid bone loss | At surgery
  Comparaison of the glenoid bone loss between both group
Surgical time | At surgery
  Comparaison og the surgery time between both group
Blood test | Before surgery
  Evaluation of the glenoid quality with nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Rouleau, MD, Principal Investigator — Université de Montréal
Locations (1):
- Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec, Canada